CLINICAL TRIAL: NCT00021151
Title: CAMPATH-1H Compassionate Treatment In Patients With PLL Who Have Failed At Least One Prior Regimen And CLL Patients Who Have Failed Fludarabine Therapy
Brief Title: Compassionate Use of Campath-1H in Treating Patients With Refractory Prolymphocytic Leukemia or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILEX1999; CWRU-ILEX-1999; ILEX-CAM511-A1; NCI-G01-1977
Record Dates: First submitted 2001-07-11; First posted 2004-04-13 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Leukemia
Keywords: refractory chronic lymphocytic leukemia; prolymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab (Experimental)
  Interventions: Biological: alemtuzumab

INTERVENTIONS:
Biological: alemtuzumab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Compassionate use refers to providing a drug to a patient on humanitarian grounds before the drug has received official approval.

PURPOSE: Compassionate use of Campath-1H in treating patients who have refractory prolymphocytic leukemia or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Expand access to Campath-1H for patients with refractory prolymphocytic leukemia or chronic lymphocytic leukemia.

OUTLINE: Patients receive Campath-1H IV over 2 hours on days 1, 3, and 5. Treatment repeats weekly for 4-12 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS: Confirmed prolymphocytic leukemia (PLL) or chronic lymphocytic leukemia (CLL) PLL that has failed at least 1 prior regimen CLL that has failed prior fludarabine, defined as: No response Disease progression while receiving therapy OR Relapse within 6 months of completion of last dose

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) (unless secondary to direct liver infiltration with CLL) Renal: Creatinine no greater than 2 times ULN Other: HIV negative No active infection No other severe concurrent disease No mental disorders No prior allergic reaction to rat or mouse-derived CDR-grafted humanized monoclonal antibodies Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy No concurrent cytotoxic therapy Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2000-01; Primary Completion 2001-04 (Actual); Study Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard J. Silver, MD, Study Chair — University Hospitals Seidman Cancer Center
Locations (1):
- Ireland Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Keating MJ, Flinn I, Jain V, Binet JL, Hillmen P, Byrd J, Albitar M, Brettman L, Santabarbara P, Wacker B, Rai KR. Therapeutic role of alemtuzumab (Campath-1H) in patients who have failed fludarabine: results of a large international study. Blood. 2002 May 15;99(10):3554-61. doi: 10.1182/blood.v99.10.3554. PMID 11986207